CLINICAL TRIAL: NCT04113005
Title: Safety and Tolerability Analysis of Combining Desmopressin With Docetaxel for the Treatment of Castration-Resistant Prostate Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Desmopressin Trial
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Castrate Resistance Prostate Cancer
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Intervention Model Description: Safety and Tolerability Analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Desmopressin (Experimental): Aim to evaluate the safety and tolerability of Desmopressin in CRPC subjects starting Docetaxel treatment.
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — To evaluate the safety and tolerability of Desmopressin in CRPC subjects starting Docetaxel treatment. Additionally, CTCs will be collected before and after Desmopressin/Docetaxel treatment to evaluate therapeutic efficacy.

SUMMARY:
This is a single site, prospective, Phase 1 pilot trial intended to evaluate the safety and tolerability of adding one IV dose of Desmopressin to CRPC subjects at least 30 minutes prior to commencing standard IV Docetaxel treatment7,8.

DETAILED DESCRIPTION:
Following Desmopressin/Docetaxel treatment subjects will be subjected to routine medical oncology follow-up, including clinical appointments, laboratory and imaging workup as well as additional Docetaxel therapy every 21 days as indicated.

An additional study clinical appointment with blood work will be organized two days post Desmopressin/Docetaxel treatment. Furthermore, for detailed documentation of AEs during the first 21 days following Desmopressin/Docetaxel therapy, subjects will be assessed weekly via phone, and in person by the investigator/treating medical oncologist before the second dose of docetaxel.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible for inclusion in this study only if all of the following criteria apply:

1. Men over 18 years of age with histologically confirmed adenocarcinoma of the prostate.
2. Signed Informed Consent Form indicating that the subject understands the purpose of, and procedures required for, the study and is willing to participate in the study.
3. Castration-resistant stage of disease about to be treated with Docetaxel.
4. Baseline laboratory values as stated below:

   1. Absolute neutrophil count ≥1.5 x 109/L;
   2. Platelet count ≥125 x 109/L;
   3. Creatinine ≤1.5 x upper limit of normal;
   4. Urea ≤1.5 x upper limit of normal;
   5. Bilirubin ≤1.1 x upper limit of normal (unless elevated secondary to conditions such as Gilbert's disease);
   6. Aspartate transaminase (AST) ≤1.5 x upper limit of normal;
   7. Alanine transaminase (ALT) ≤1.5 x upper limit of normal;
   8. Castrate serum testosterone level (< 1.7 nmol/L).

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Known Desmopressin intolerability.
2. Any state of known congestive heart disease (CHF class >1).
3. Sodium blood levels < 135 mEq/ml at enrollment.
4. Eastern Cooperative Oncology Group (ECOG) performance status >1.
5. Moderate or severe chronic kidney disease (eGFR <60 mL/min).
6. Prior use of docetaxel for CRPC.
7. ≤30 days prior to study treatment received or had:

   1. Transfusion (platelets or red blood cells), or hematopoetic growth factors;
   2. Any type of chemotherapy;
   3. Any form of hormonal treatment with the exception of the continuous GnRH analogues required to maintain castrate state;
   4. Corticosteroid treatment equivalent to >10 mg of Prednisone orally daily;
   5. An investigational agent for prostate cancer;
   6. Ongoing Desmopressin therapy at enrollment;
   7. Major surgery.
8. Current use of: Clofibrate, Chlorpropamide, Carbamazepine, Demeclocycline, Lithium, or Norepinephrine.
9. History of or current documented brain metastasis or carcinomatous meningitis, treated or untreated (brain imaging for asymptomatic subjects is not required).
10. Current symptomatic cord compression requiring surgery or radiation therapy (once successfully treated and there has been no progression, subjects are eligible for the study).
11. Uncontrolled medical conditions such as diabetes mellitus, angina pectoris, serious cardiac arrhythmia, severe hypertension, or active infection requiring systemic antibiotics, or any event such as myocardial infarction, cerebrovascular accident, or pulmonary embolism within 3 months prior to protocol therapy, as well as any significant concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects presenting with AEs within a 21-day period of time post Desmopressin/Docetaxel treatment; nature and severity of AEs (as per Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, Appendix B). | 12 months
  Number of subjects presenting with AEs within a 21-day period of time post Desmopressin/Docetaxel treatment; nature and severity of AEs (as per Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, Appendix B).
  The proportion of subjects presenting with hyponatremia at 48-hour time point; severity of hyponatremia as per CTCAE Version 4.03 (Appendix B).

CONTACTS AND LOCATIONS:
Overall Officials: Urban Emmenegger, Principal Investigator — Sunnybrook Research Institute

IPD SHARING:
Plan to Share IPD: No